CLINICAL TRIAL: NCT01708291
Title: HEALTHY (Health Education Adolescent Leadership Training to Help Youth) Leaders
Acronym: HEALTHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Sandra Jee, Associate Professor of Pediatrics, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PMA 2-12213
Record Dates: First submitted 2012-09-04; First posted 2012-10-16 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Stress
Keywords: youth; Stress; mindfulness; foster care; stress reduction; high risk teens
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Stress reduction (Active Comparator): attending 10 weekly sessions and comprised of an eight week mindfulness intervention program, and completing pre- and postevaluation measures on the first and last sessions
  Interventions: Behavioral: Mindfulness based stress reduction
- No Mindfulness based intervention (Placebo Comparator): completing only re- and post-evaluation measures on the first and last sessions
  Interventions: Behavioral: only pre and post evaluation measures

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — an 8 week group intervention to teach mindfulness skills
  Arms: Mindfulness Based Stress reduction
Behavioral: only pre and post evaluation measures
  Arms: No Mindfulness based intervention

SUMMARY:
This project will measure baseline stress among a group of youth in foster and kinship care. The investigators will implement a pilot program to target stress reduction by using an evidence-based group therapy technique teaching mindfulness skills. The investigators hypothesize that the mindfulness skills will help youth to reduce stress, which will be measured using psychological and physiological techniques.

ELIGIBILITY:
Inclusion Criteria:

* ages 14-21 years at time of intervention being offered, offered to youth in out of home care (e.g. foster and kinship care)

Exclusion Criteria:

* severe developmental delay
* non English speaking, not in age range

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Jee SH, Szilagyi M, Conn AM, Nilsen W, Toth S, Baldwin CD, Szilagyi PG. Validating office-based screening for psychosocial strengths and difficulties among youths in foster care. Pediatrics. 2011 May;127(5):904-10. doi: 10.1542/peds.2010-1350. Epub 2011 Apr 18. PMID 21502256
- [Background] Jee SH, Halterman JS, Szilagyi M, Conn AM, Alpert-Gillis L, Szilagyi PG. Use of a brief standardized screening instrument in a primary care setting to enhance detection of social-emotional problems among youth in foster care. Acad Pediatr. 2011 Sep-Oct;11(5):409-13. doi: 10.1016/j.acap.2011.03.001. Epub 2011 Jun 17. PMID 21683668
- [Derived] Jee SH, Couderc JP, Swanson D, Gallegos A, Hilliard C, Blumkin A, Cunningham K, Heinert S. A pilot randomized trial teaching mindfulness-based stress reduction to traumatized youth in foster care. Complement Ther Clin Pract. 2015 Aug;21(3):201-9. doi: 10.1016/j.ctcp.2015.06.007. Epub 2015 Jun 20. PMID 26256140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were not included in the study due to fighting.
Groups:
- Mindfulness Based Stress Reduction: Will complete 10 weekly sessions and comprised of an 8 week mindfulness intervention program and completing pre- and post-evaluation measures on the first and last sessions.
- No Mindfulness Based Stress Reduction: Will complete pre and post evaluation measures on the first and last sessions with no weekly sessions or mindfulness intervention program.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | No Mindfulness Based Stress Reduction
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1
Not completed — fighting | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for 3 subjects. They were excluded from the study for fighting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | No Mindfulness Based Stress Reduction | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Customized [Number; unit: participants]
  14 to 17 | 17 | 5 | 22
  18 to 21 | 4 | 16 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 15 | 31
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Pediatric Symptoms as Assessed by the Pediatric Symptom Checklist-17 (PSC-17)
Description: Self Administered questionnaire to assess level of stress at baseline and week 10. PSC-17 is a one page behavioral assessment tool that can be completed in <5 minutes and can assess the sub-domains of attention, externalizing problem and internalizing problems. Attention, externalizing and Internalizing domains are each scored on a scale from 0 (best) to 10 (worst), where a score >= 7 indicates stress.
Time Frame: Baseline and week 10
Measure: Number; unit: participants
Arm/Group | Mindfulness Based Stress Reduction | No Mindfulness Based Stress Reduction
Number analyzed (Participants) | 21 | 21
participants
  week 0-attention | 3 | 2
  week 0-external | 4 | 3
  week 0-internal | 4 | 8
  week 10-attention | 3 | 4
  week 10-external | 3 | 3
  week 10-internal | 6 | 11

ADVERSE EVENTS:
Arm/Group | Mindfulness Based Stress Reduction | No Mindfulness Based Stress Reduction
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes